CLINICAL TRIAL: NCT04605445
Title: One Vs Two Visits Endodontics - a Prospective Randomized Multicenter Study in General Dental Practice
Brief Title: One Vs Two Visits Root Canal Treatments in Infected Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Collaborators: Norrbottens County Council (Other Government); Landstinget i Kalmar Län (Other); Blekinge County Council (Unknown); Kronoberg County Council (Other Government); Odontologisk Forskning i Region Skåne (OFRS) (Unknown); County Council of Halland, Sweden (Other Government); Smile Tandvård (Unknown); Aragón Dental (Unknown); Kalmar County Council (Unknown); Oris Dental (Unknown)
Responsible Party: Principal Investigator, Annika E Björkner, Associate Professor, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPN 2020-00207
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Apical Periodontitis; Pain; Tooth Loss; Dental Pulp Necrosis
Keywords: Endodontics; General Dental Practice; Single Visit; Multiple Visits; Infection Barrier
MeSH Terms: conditions — Periapical Periodontitis; Pain; Tooth Loss; Dental Pulp Necrosis | interventions — Endodontics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 visit endodontics (Experimental): Root canal treatment is performed in one visit.
  Interventions: Procedure: 1 visit root canal treatment (endodontics)
- 2 visits endodontics (Active Comparator): Root canal treatment is performed in two visits.
  Interventions: Procedure: 2 visits root canal treatment (endodontics)

INTERVENTIONS:
Procedure: 1 visit root canal treatment (endodontics) — Endodontics (root canal treatment). In the enrolment visit, access, opening and identification of root canals can be performed and a suitable temporization will be placed in the tooth if needed. Root canal treatment can be completed in the same visit or performed in another visit where cleaning, shaping and root filling procedures, temporization or permanent restoration will be performed. These procedures are part of the normal clinical praxis. No rigid protocol will be implemented, as a pragmatic design was chosen.
  Arms: 1 visit endodontics
Procedure: 2 visits root canal treatment (endodontics) — Endodontics (root canal treatment). In the enrolment visit, access, opening and identification of root canals can be performed and a suitable temporization will be placed in the tooth if needed. Root canal treatment can be started, or performed in another visit, lasting 2 visits. In the first visit cleaning and shaping is performed and a medication is put in place in the canals, and the tooth is temporized until the next visit at least one week apart. In the second visit the tooth is root filled and temporization or permanent restoration will be performed. These procedures are part of the normal clinical praxis. No rigid protocol will be implemented, as a pragmatic design was chosen.
  Arms: 2 visits endodontics

SUMMARY:
The primary aim of the study is to compare the outcome of one vs two visits endodontics (root canal treatments) performed in general dental practice of infected (necrotic) teeth, one and four years after treatment. Secondary aims are to compare the root filling quality and the frequency of complications for both treatment modalities.

A pilot study will identify the shortcomings of the protocol, which will be revised accordingly.

A multi-center study in several clinics from five counties throughout Sweden is planned. Consecutive eligible patients (see inclusion and exclusion criteria) with one tooth each will be included.

The study sample size calculation was based on a judgement that a minimal worthwhile effect of less than 10% was not clinically relevant. The presumption was that successful outcomes would be of 75% and 65% for the different treatment arms, respectively. Three hundred and fifty six patients per group are thus needed to detect that difference as statistical significant with a power of 80% and an alfa-error of 5%. To compensate for around 30% drop-outs a number of 1000 patients will be recruited.

Patients will be randomly enrolled in two arms: one in which the endodontic treatment (root canal treatment) is performed in one visit, and in the other arm in two visits. The allocation sequences for one vs multiple visit endodontics will be computer generated followed by a dark colored envelope concealed allocation.

The patients will be contacted by telephone 5-7 days post-operatively, and a control visit at the clinic will be scheduled one month post-operatively to assess complications related to the treatment.

A clinical control will be performed at the clinic one and four years after treatment. Intra-oral radiographs will be taken. The radiographs will be examined by two blinded and independent observers. A successful outcome is defined by clinical and radiographic normalcy.

The statistical methods selected to analyse the primary outcome will be the Chi square test of 2x2 tables, or Fisher´s exact test when proportions are small and the expected value <5. The calculations will be two-tailed. Results will be considered statistically significant at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 17 years.
* Permanent tooth excluding third molars.
* Necrotic tooth with/without clinical and/or radiological signs of apical (juxta radicular) periodontitis (non-bleeding pulp in the canal orifice. In case of a multi rooted tooth, a non-bleeding pulp in at least one root canal orifice) where orthograde endodontic treatment is planned.

Exclusion Criteria:

* Patients with severe general disease and/ or where endodontic treatment requires special consideration for health reasons (eg radiation-treated jaw bone in the area or increased susceptibility to infection).
* Systemic involvement (fever).
* Swelling (extra- and/or intra oral).
* Previously root canal treated tooth (instrumented and/or rotfilled).
* Confirmed or strong suspicion of transverse or longitudinal root fracture.
* Trauma to the tooth (<6 month).
* Marginal bone loss >1/3 of the root lenght.
* Root resorption.
* Non restorable tooth.
* Endodontic treatment is not considered feasible because rubberdam cannot be used on the tooth.
* Follow-up at the clinic of the treatment after> 1 year is considered not feasible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Periapical health at year 1 | One year after completed treatment
  Assessment of apical radio-anatomical structures by two independent and blinded observers
Periapical health at year 4 | Four years after completed treatment
  Assessment of apical radio-anatomical structures by two independent and blinded observers

SECONDARY OUTCOMES:
Post-operative pain 7 days | 5-7 days post-operatively
  Patient self-reported pain at an numeric rating scale from 0 (no pain) to 10 (worst pain imaginable)
Post-operative pain 30 days | 30 days post-operatively
  Patient self-reported pain at an numeric rating scale from 0 (no pain) to 10 (worst pain imaginable)
Medication intake | 30 days post-operatively
  Patient self-reported analgesic and antibiotic intake
Tooth survival at year 1 | 1 year after completed treatment
  Presence of root-filled tooth
Tooth survival at year 4 | 4 year after completed treatment
  Presence of root-filled tooth
Complications | 30 days and long-term follow-up at year 1 and 4
  Complications not previously described that can be associated with endodontic treatment

CONTACTS AND LOCATIONS:
Locations (7):
- Sweden (7):
  - Folktandvården Region Kronoberg, Vaxjo, Kronoberg County
  - Folktandvården Region Norrbotten, Luleå, Norrbotten County
  - Folktandvården Region Kalmar, Kalmar
  - Smile Tandvård, Luleå
  - Aragón Dental, Malmo
  - Oris Dental, Malmo
  - Folktandvården Region Halland, Varberg

IPD SHARING:
Plan to Share IPD: No